CLINICAL TRIAL: NCT01538628
Title: Evaluation of SpaceOAR™ System When Used to Create Space Between the Rectum and Prostate in Men Undergoing IG-IMRT for Localized Stage T1-T2 Prostate Cancer: A Randomized, Multicenter, Parallel Arm Controlled Clinical Study
Brief Title: SpaceOAR System Pivotal Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Augmenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGX-11-001-US
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Spacer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SpaceOAR (Experimental): Men meeting the study eligibility criteria will be scheduled for fiducial marker placement using a transperineal approach with ultrasound guidance. Following successful fiducial marker placement, subjects will be randomized (2:1) to the treatment group or control group. Subjects randomized to the treatment group will undergo placement of 10 mL of SpaceOAR hydrogel
  Interventions: Device: SpaceOAR System
- Control (No Intervention): Men meeting the study eligibility criteria will be scheduled for fiducial marker placement using a transperineal approach with ultrasound guidance. Following successful fiducial marker placement, subjects will be randomized (2:1) to the treatment group or control group. Subjects randomized to the control group will not receive injection of the SpaceOAR hydrogel.

INTERVENTIONS:
Device: SpaceOAR System — Fiducial marker placement followed by randomization to treatment group, i.e., 10mL SpaceOAR hydrogel injection, or control group, i.e., no injection of SpaceOAR hydrogel.
  Arms: SpaceOAR

SUMMARY:
Evaluate the safety of the SpaceOAR System when the hydrogel is injected between the rectum and prostate in men undergoing radiation therapy (IG-IMRT)

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of the SpaceOAR System when the hydrogel is injected between the rectum and prostate in men undergoing radiation therapy (IG-IMRT) and to evaluate whether use of the SpaceOAR hydrogel results in a reduction of radiation exposure to the anterior rectum.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than 18 years old
* Subjects must have pathologically confirmed invasive adenocarcinoma of the prostate and must be planning to undergo IMRT
* Subjects must have clinical stage T1 or T2 as determined from a biopsy taken within 6 months of the baseline/screening visit with Gleason Score less than or equal to 7
* Subjects Screening/Baseline laboratory testing must meet the following laboratory value criteria: PSA less than or equal to 20 ng/mL,hematocrit greater than 30%,serum creatinine less than 2.0 mg/dl, serum AST and ALT less than 2.5 times upper limit of institution normal, and serum bilirubin less than 2.0 mg/dl
* Subject or authorized representative, has been informed of the nature of the study and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site

Exclusion Criteria:

* Prostate greater than 80cc documented within 3 months preceding the Screening/Baseline visit
* Subjects with extracapsular extension of the prostate cancer, with greater than 50% of the number of biopsy cores positive for cancer, metastatic disease, other ongoing cancers which will be treated during the study, or subjects for whom pelvic lymph node radiotherapy is planned
* Subjects with any prior invasive malignancy (except non-melanomatous skin cancer) unless the subject has been disease free for a minimum of 5 years.
* Subjects who are indicated for androgen deprivation therapy or who have been treated with androgen therapy within the prior 3 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Urological Surgeons of Northern California, Campbell, California
  - Radiological Associates of Sacramento, Sacramento, California
  - The Urology Center of Colorado, Denver, Colorado
  - Lakewood Ranch Oncology Center/21st Century Oncology, Bradenton, Florida
  - 21st Century Oncology, Fort Myers, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University Department of Radiation Oncology and Molecular Radiation Sciences, Baltimore, Maryland
  - Chesapeake Urology Associates, Chesapeake Urology Research Associates (The Prostate Center), Owings Mills, Maryland
  - Northern Nevada Radiation Oncology, Reno, Nevada
  - CentraState Medical Center, Freehold, New Jersey
  - Western New York Urology Associates, LLC and D/B/A Cancer Care of WNY, Erie, Niagara, and Chautauqua County, New York
  - Advanced Radiation Centers of New York, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - Upstate Medical University, Syracuse, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - 21st Century Oncology, Myrtle Beach, South Carolina
  - Peninsula Cancer Center, Poulsbo, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was treated on January 27, 2012 and the last subject visit occurred on July 15, 2014.
Pre-assignment Details: Randomized study, no wash out or run-in period
Groups:
- SpaceOAR: Subjects meeting the study eligibility criteria will be scheduled for fiducial marker placement using a transperineal approach with ultrasound guidance. Following successful fiducial marker placement, subjects will be randomized (2:1) to the treatment group or control group. Subjects randomized to the treatment group will undergo placement of 10 mL of SpaceOAR hydrogel
  SpaceOAR System: Fiducial marker placement followed by randomization to treatment group, i.e., 10mL SpaceOAR hydrogel injection, or control group, i.e., no injection of SpaceOAR hydrogel.
- Control: Subjects meeting the study eligibility criteria will be scheduled for fiducial marker placement using a transperineal approach with ultrasound guidance. Following successful fiducial marker placement, subjects will be randomized (2:1) to the treatment group or control group. Subjects randomized to the control group will not receive injection of the SpaceOAR hydrogel.
Period: Overall Study
Arm/Group | SpaceOAR | Control
Started | 149 | 73
Completed | 148 | 71
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SpaceOAR: Subjects randomized to receive SpaceOAR hydrogel.
- Control: Subjects randomized to not receive SpaceOAR hydrogel.
- Total: Total of all reporting groups
Arm/Group | SpaceOAR | Control | Total
Number analyzed (Participants) | 149 | 73 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.36 (7.73) | 67.66 (6.51) | 66.39 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 149 | 73 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 144 | 71 | 215
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Subjects may check more than one category, therefore this is why SpaceOAR subjects = 150/149.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 16 | 8 | 24
    White | 127 | 61 | 188
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 149 | 73 | 222

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving a Reduction of 25% or Greater in Percent Volume of the Rectum Receiving at Least 70 Gy Measured From CT Scans Acquired Pre and Post SpaceOAR Hydrogel Injection
Description: Measurements calculated and documented by the Core Lab. Measurements performed with the Core Lab blinded to subject identification. Results based on the Core Lab computation are considered as primary.
Time Frame: 3 months post index procedure
Population: SpaceOAR Group Only
Measure: Count of Participants; unit: Participants
Arm/Group | SpaceOAR
Number analyzed (Participants) | 147
Participants | 143
Statistical Analysis 1: Comparison: SpaceOAR; Test type: Superiority or Other; p = .0001, Exact binomial test; testing the null hypothesis that the proportion for SpaceOAR is less than or equal to 0.70

2. Primary Outcome: Percentage of Subjects Experiencing Grade 1 or Greater Rectal or Procedure Adverse Events Post Index Procedure
Description: The primary safety endpoint was the occurrence of Grade 1 or greater rectal adverse events or procedure adverse events in the 6 months following the Index Procedure. The numbers reflect the percent of subjects in each arm/group that experienced grade 1 or greater rectal or procedure adverse events post index procedure.
Time Frame: 6 months post index procedure
Population: Intent-to-Treat (ITT) population was defined to be all randomized subjects (SpaceOAR and Control group).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | SpaceOAR | Control
Number analyzed (Participants) | 149 | 73
percentage of subjects | 34.2 [26.7 to 42.4] | 31.5 [21.1 to 43.4]

3. Secondary Outcome: Percentage of Subjects Experiencing Grade 2 or Greater Rectal or Procedure Adverse Events in the 6 Months Following the Index Procedure
Description: The numbers reflect the percent of subjects in each arm/group that experienced grade 2 or greater rectal or procedure adverse events post index procedure.
Time Frame: 6 months post index procedure
Population: Intent-to-Treat (ITT) population was defined to be all randomized subjects (SpaceOAR and Control group).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | SpaceOAR | Control
Number analyzed (Participants) | 149 | 73
percentage of subjects | 10 [3.3 to 12.0] | 3 [0.9 to 11.5]

4. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite (EPIC) Score Following Index Procedure
Description: Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive survey instrument designed to assesses the disease-specific aspects of prostate cancer and its therapies and comprises four domains. Scores for each domain (urinary, sexual, bowel, hormonal) range from 0-100, with higher scores indicating improved quality of life. Scores are reported as mean change from baseline at each time point.
Time Frame: 3 months, 6 months, 12 months, 15 months
Population: Intent-to-Treat (ITT) population was defined to be all randomized subjects (SpaceOAR and Control group). Mean change in score was calculated for the number of subjects providing data at each follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SpaceOAR | Control
Number analyzed (Participants) | 149 | 73
score on a scale
  Change in Urinary Assessment Composite Score at 3 Months: number analyzed (Participants) | 146 | 65
  Change in Urinary Assessment Composite Score at 3 Months | -11.69 (13.20) | -11.20 (16.50)
  Change in Urinary Assessment Composite Score at 6 Months: number analyzed (Participants) | 144 | 71
  Change in Urinary Assessment Composite Score at 6 Months | 1.38 (9.82) | -0.83 (13.12)
  Change in Urinary Assessment Composite Score at 12 Months: number analyzed (Participants) | 142 | 70
  Change in Urinary Assessment Composite Score at 12 Months | 0.12 (11.74) | 0.30 (13.51)
  Change in Urinary Assessment Composite Score at 15 Months: number analyzed (Participants) | 144 | 68
  Change in Urinary Assessment Composite Score at 15 Months | 1.69 (11.74) | 2.2 (11.66)
  Change in Sexual Assessment Composite Score at 3 Months: number analyzed (Participants) | 140 | 64
  Change in Sexual Assessment Composite Score at 3 Months | -7.60 (17.36) | -4.86 (19.83)
  Change in Sexual Assessment Composite Score at 6 Months: number analyzed (Participants) | 137 | 69
  Change in Sexual Assessment Composite Score at 6 Months | -3.44 (16.74) | -2.35 (18.68)
  Change in Sexual Assessment Composite Score at 12 Months: number analyzed (Participants) | 138 | 68
  Change in Sexual Assessment Composite Score at 12 Months | -7.21 (19.32) | -8.29 (20.51)
  Change in Sexual Assessment Composite Score at 15 Months: number analyzed (Participants) | 137 | 66
  Change in Sexual Assessment Composite Score at 15 Months | -6.55 (19.71) | -5.33 (21.52)
  Change in Bowel Habits Assessment Composite Score at 3 Months: number analyzed (Participants) | 145 | 65
  Change in Bowel Habits Assessment Composite Score at 3 Months | -7.47 (12.69) | -6.24 (12.05)
  Change in Bowel Habits Assessment Composite Score at 6 Months: number analyzed (Participants) | 143 | 68
  Change in Bowel Habits Assessment Composite Score at 6 Months | -0.78 (8.52) | -2.44 (9.54)
  Change in Bowel Habits Assessment Composite Score at 12 Months: number analyzed (Participants) | 142 | 69
  Change in Bowel Habits Assessment Composite Score at 12 Months | -0.95 (9.69) | -3.08 (8.61)
  Change in Bowel Habits Assessment Composite Score at 15 Months: number analyzed (Participants) | 143 | 66
  Change in Bowel Habits Assessment Composite Score at 15 Months | -0.02 (9.41) | -2.14 (9.29)
  Change in Hormonal Assessment Composite Score at 3 Months: number analyzed (Participants) | 141 | 61
  Change in Hormonal Assessment Composite Score at 3 Months | -2.69 (9.96) | -3.87 (8.99)
  Change in Hormonal Assessment Composite Score at 6 Months: number analyzed (Participants) | 139 | 67
  Change in Hormonal Assessment Composite Score at 6 Months | -0.71 (9.05) | -2.35 (11.33)
  Change in Hormonal Assessment Composite Score at 12 Months: number analyzed (Participants) | 135 | 65
  Change in Hormonal Assessment Composite Score at 12 Months | -0.71 (9.45) | -0.81 (8.88)
  Change in Hormonal Assessment Composite Score at 15 Months: number analyzed (Participants) | 137 | 65
  Change in Hormonal Assessment Composite Score at 15 Months | 0.03 (9.58) | 0.70 (8.92)

5. Secondary Outcome: Percentage of Subjects Requiring at Least One Medication Change for Mitigation of Rectal or Urinary Symptoms or for Procedure-related Events in the 6 Months Following the Index Procedure
Description: The numbers reflect the percent of subjects in each arm/group that required at least one medication change to treat rectal or urinary symptoms in the 6 months post index procedure.
Time Frame: 6 months post procedure
Population: Intent-to-Treat (ITT) population was defined to be all randomized subjects (SpaceOAR and Control group).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | SpaceOAR | Control
Number analyzed (Participants) | 149 | 72
percentage of subjects | 56.4 [48.0 to 64.5] | 63.9 [51.7 to 74.9]

6. Secondary Outcome: Number of SpaceOAR Subjects Experiencing a Procedure-Related Adverse Event (AE) Prior to Initiation of Radiation Therapy
Description: An event was classified as a Procedure AE if it occurred during during and immediately after the Index Procedure or was deemed to be associated with the Index Procedure by the Clinical Events Committee (CEC). Per protocol subjects were to begin intensity modulated radiation therapy within 21 days following fiducial marker and/or SpaceOAR placement.
Time Frame: 21 days post index procedure, prior to initiation of radiation therapy
Population: SpaceOAR treated subjects experiencing a procedure related AE prior to initiation of radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | SpaceOAR
Number analyzed (Participants) | 149
Participants | 14

7. Secondary Outcome: Number of Subjects Experiencing a Delay in Radiation Therapy Associated With a Procedure or Device-Related Adverse Event
Description: All subjects begin Intensity Modulated Radiation Therapy (IMRT) within 21 days following index procedure (Fiducial Marker Placement with or without SpaceOAR Hydrogel Injection).
Time Frame: 21 days post index procedure
Population: Intent-to-Treat (ITT) population was defined to be all randomized subjects (SpaceOAR and Control group).
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | SpaceOAR | Control
Number analyzed (Participants) | 149 | 73
participants | 0 [0.0 to 2.4] | 0 [0.0 to 4.9]

ADVERSE EVENTS:
Arm/Group | SpaceOAR | Control
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/73
Serious Adverse Events (participants affected / at risk) | 21/149 | 10/73
Other Adverse Events (participants affected / at risk) | 17/149 | 2/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SpaceOAR (N=149) | Control (N=73)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Corneal dystrophy (Eye disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Renal cell carcinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SpaceOAR (N=149) | Control (N=73)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anorectal pressure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Discomfort while sitting (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal penetration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vasovagal presyncope (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No